CLINICAL TRIAL: NCT00383734
Title: Randomized, Comparative, Multicenter, Patient-blinded Trial of the Safety and Efficacy of Intradermal Injections of Polylactic Acid (Newfill TM) Versus Polyacrylamid Gel (Eutrophill) in the Treatment of Facial Lipoatrophy in HIV-infected Patients ANRS 132 SMILE
Brief Title: Safety and Efficacy of Intradermal Injections of Newfill Versus Eutrophill in the Treatment of Facial Lipoatrophy in HIV-infected Patients ANRS 132 SMILE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Procitech (Unknown); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANRS 132
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV-Associated Lipodystrophy Syndrome
Keywords: HIV-Associated Lipodystrophy Syndrome; polylactic acid; polyacrylamide gels
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): newfill
  Interventions: Device: Newfill
- 2 (Experimental): Eutrophill
  Interventions: Device: Eutrophill

INTERVENTIONS:
Device: Newfill — 1 to 7 injections of drug
  Arms: 1
Device: Eutrophill — 1 to 7 injections of drug
  Arms: 2

SUMMARY:
Treatment of facial lipoatrophy with dermal injections polylactic acid (Newfill TM) is a safe procedure and has been now widely used with a good efficacy. However, this therapy is not effective in all treated patients and the benefit of the injections may decrease with time necessitating re-injections several months after the first sets of injections. In this study we would like to compare the efficacy and safety of Eutrophill(polyacrylamid gel), a resorbable filler compound versus Newfill in a comparative, randomised, multicenter trial. Primary endpoint will be the self-perception by the patient with a visual analogue scale (VAS index). Secondary endpoints are a quality of life questionnaire (MOS-HIV), the a-NBC questionnaire (perception by the patient and by the doctor of the severity of the lipoatrophy), the measure of the dermal thickness and cheek skin fold as assessed by the Skinfold Caliper, the ordering of digital photographs and the evaluation of the dermal thickness by CT scan.

DETAILED DESCRIPTION:
The aim of the study is to compare the efficacy and safety of Eutrophill (polyacrylamid gel), a resorbable filler compound versus Newfill( polylactic acid) in a comparative, randomised, multicenter trial and patient-blinded study, in the treatment of facial lipoatrophy in HIV-infected patients, one year after the first injection (week 48). The efficacy will be assessed by measuring the median self-perception index of the patients with a visual analogue scale (VAS index).The study will compare between treatments, at week 48, week 72 and week 96 versus baseline :the median increase of the VAS index, the rate of treatment failure, the scores of 2 patients-questionnaires (a-NBC and MOS-HIV),the ordering of digital photographs,the median increase of the facial dermal thickness of the cheek and the dermal skin fold as assessed by a Skinfold Caliper.

The study will compare at week 48 and week 96 versus baseline:

the median increase of dermal thickness as assessed by CT scan of the face. Safety will be assessed by the frequency and nature of immediate and delayed side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* confirmed laboratory diagnosis of HIV infection
* facial lipoatrophy
* stable antiretroviral treatment or no treatment for at least 3 months
* written informed consent

Exclusion Criteria:

* history of surgical or cosmetic intervention for facial lipoatrophy
* no history of antiretroviral therapy
* current opportunistic infection
* currently stavudine containing antiretroviral regimen
* CD4 cell count under 200per µL, plasma HIV RNA above 10000 copies per mL under antiretroviral therapy
* platelets under 50000 per µL and or abnormal coagulation tests
* pregnancy
* major or concomitant illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
- patient's subjective self-perception of improvement of facial lipoatrophy as assessed by a VAS | week 48

SECONDARY OUTCOMES:
quality of life questionnaire,NBC questionnaire, dermal thickness and cheek skin fold as assessed by the Skinfold Caliper, digital photographs, dermal thickness as assessed by CT scan | week 0, week 48 and week 96

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Lafaurie, MD, Principal Investigator — Hopital Saint Louis AP-HP; Raphael Porcher, MD, Study Chair — Hôpital Saint-Louis AP-HP
Locations (1):
- Hôpital Saint-Louis Service des Maladies Infectieuses, Paris, France

REFERENCES:
- [Derived] Lafaurie M, Dolivo M, Girard PM, May T, Bouchaud O, Carbonnel E, Madelaine I, Loze B, Porcher R, Molina JM; ANRS 132 SMILE study group. Polylactic acid vs. polyacrylamide hydrogel for treatment of facial lipoatrophy: a randomized controlled trial [Agence Nationale de Recherches sur le SIDA et les Hepatites Virales (ANRS) 132 SMILE]. HIV Med. 2013 Aug;14(7):410-20. doi: 10.1111/hiv.12021. Epub 2013 Feb 24. PMID 23432777